CLINICAL TRIAL: NCT04245865
Title: Tocotrienol and Bevacizumab in Metastatic Colorectal Cancer. A Randomized Phase II Marker Trial
Brief Title: Tocotrienol and Bevacizumab in Metastatic Colorectal Cancer
Acronym: Toco-CoR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Toco-CoR
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal cancer; Tocotrienol; Natural killer cells; Circulating tumor DNA
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Bevacizumab; Capecitabine; Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A, standard treatment + tocotrienol (Experimental): Fluorouracil + calcium folinate + oxaliplatin + bevacizumab + tocotrienol OR capecitabine + bevacizumab + tocotrienol
  Interventions: Drug: Fluorouracil; Drug: Calcium folinate; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine; Dietary Supplement: Tocotrienol
- Arm B, standard treatment + placebo (Placebo Comparator): Fluorouracil + calcium folinate + oxaliplatin + bevacizumab + placebo OR capecitabine + bevacizumab + placebo
  Interventions: Drug: Fluorouracil; Drug: Calcium folinate; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine; Other: Placebo

INTERVENTIONS:
Drug: Fluorouracil — 2800 mg/m2 iv
Drug: Calcium folinate — 400 mg/m2 iv
Drug: Oxaliplatin — 85 mg/m2 iv
Drug: Bevacizumab — 5 mg/kg OR 7.5 mg/kg iv
Drug: Capecitabine — 2000 mg/m2 orally daily for two weeks
Dietary Supplement: Tocotrienol — 300 mg orally x 3 daily
  Arms: Arm A, standard treatment + tocotrienol
Other: Placebo — Placebo orally x 3 daily
  Arms: Arm B, standard treatment + placebo

SUMMARY:
This double blind, randomized phase II trial will investigate whether the addition of tocotrienol will improve the effect and lower the toxicity of standard chemotherapy and bevacizumab. Half of the patients will receive tocotrienol and the other half placebo. Treatment is planned for a period of maximum six months and will be discontinued earlier in case of progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified adenocarcinoma of the colon or rectum
* Metastatic disease
* Planned treatment with FOLFOX or capecitabine combined with bevacizumab
* Evaluable disease according to RECIST 1.1
* Performance status 0-2
* Expected survival ≥ 3 months
* Patient acceptance to collection of blood samples for translational research
* Age ≥ 18 years
* Contraception during and 6 months after last dose for women of childbearing potential (less than one year amenorrhea and not undergone hysterectomy, bilateral salpingectomy or bilateral oophorectomy) and for male patients with a fertile partner. Hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or sexual abstinence is accepted.
* Adequate bone marrow function, liver function, and renal function (within 7 days prior to inclusion):

  * WBC ≥ 3.0 x 109/l or neutrophils (ANC) ≥ 1.5 x 10^9/l
  * Platelet count ≥ 100 x 10^9/l
  * Hemoglobin ≥ 6.0 mmol/l
  * Serum bilirubin ≤ 2.0 x ULN
  * Serum transaminase ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 ULN
* Urine dipstick for protein ≤ 2+, if the dipstick shows protein ≥ 2+, 24 hour urine testing must be performed and show protein contents ≤ 1g.
* Written and orally informed consent

Exclusion Criteria:

* Other active malignant disease within 5 years prior to inclusion in the study.
* Other experimental therapy within 28 days prior to treatment initiation.
* Underlying medical disease not adequately treated.
* Surgery, including open biopsy, within 4 weeks prior to first dose of bevacizumab.
* Cerebral vascular attack, transient ischemic attack or subarachnoid hemorrhage within six months before start of treatment
* Bleeding tumor
* Pregnant or breastfeeding women
* Fertile patients not willing to use effective methods of contraception during treatment and for six months after end of treatment.
* Hypersensitivity to one or more active substances or auxiliary substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The rate of progression free patients at six months | Six months after enrollment of the last patient

SECONDARY OUTCOMES:
Time to first serious adverse event according to CTCAE 5.0 | Six months after enrollment of the last patient
  CTCAE=Common Terminology Criteria for Adverse Events
Response rate as measured by RECIST 1.1 | Six months after enrollment of the last patient
  RECIST=Response evaluation criteria in solid tumors
Overall survival | 12 months after enrollment of the last patient

CONTACTS AND LOCATIONS:
Overall Officials: Torben F Hansen, MD, PhD, Study Chair — Department of Oncology, Vejle Hospital - University Hospital of Southern Denmark
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark